CLINICAL TRIAL: NCT00965458
Title: Inducing Remission in New Onset Type 1 Diabetes Mellitus With Alefacept (Amevive®)
Brief Title: Inducing Remission in Type 1 Diabetes With Alefacept
Acronym: T1DAL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Manufacturer discontinued production of Amevive®: business decision.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network); Juvenile Diabetes Research Foundation (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAIT ITN045AI
Record Dates: First submitted 2009-08-22; First posted 2009-08-25 (Estimated); Results first posted 2015-01-07 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-06

CONDITIONS: New-onset Type 1 Diabetes Mellitus
Keywords: New-onset Type 1 Diabetes Mellitus; New-onset T1DM; New-onset T1D; Alefacept; Amevive®
MeSH Terms: interventions — Alefacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alefacept (Experimental): Subjects in this group receive weekly intramuscular injections of alefacept (15 mg) for 2 cycles of 12 weeks each, separated by a 12 week pause in treatment.
  Interventions: Biological: Alefacept
- Placebo (Placebo Comparator): Subjects in this group received weekly intramuscular injections of a placebo saline solution of equal volume to the alefacept group for 2 cycles of 12 weeks each, separated by a 12 week pause in treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Alefacept — Weekly intramuscular injections of alefacept (15 mg) for 2 cycles of 12 weeks each, separated by a 12 week pause in treatment.
  Other Names: Amevive®
  Arms: Alefacept
Drug: Placebo — Weekly intramuscular injections of a placebo saline solution of equal volume to the alefacept group for 2 cycles of 12 weeks each, separated by a 12 week pause in treatment.
  Other Names: Inactive drug (pharmacologically)
  Arms: Placebo

SUMMARY:
The purpose of this trial is to test whether a drug called alefacept will slow or halt destruction of the beta cells in the pancreas. If the destruction of the beta cells is stopped, the patients might be able to produce insulin on their own longer, which could stop or slow the progression of their type 1 diabetes.

This is a multi-center prospective, placebo-controlled, double-blind and randomized trial to investigate the ability of alefacept to protect residual beta cells from ongoing autoimmune destruction in adolescents and young adults with newly diagnosed Type 1 Diabetes Mellitus (T1DM).

DETAILED DESCRIPTION:
T1DM is an autoimmune disease that can emerge suddenly, causing dependence on insulin for life. This means that the immune system (the part of your body that helps fight infections) mistakenly attacks the cells in the pancreas that produce insulin (beta cells). As beta cells are destroyed, one's ability to produce insulin is decreased. Insulin helps keep blood glucose (sugar) levels normal.

For a period right after diagnosis, the pancreas is still able to make small amounts of insulin. Individuals with diabetes who have the ability to produce some of their own insulin may be able to achieve better blood sugar control than people who produce no insulin at all. Based on previous research, doctors think that giving medicines to affect the immune system soon after diagnosis may stop, delay, or decrease the destruction of beta cells, resulting in better glucose control. This can help prevent secondary complications of diabetes down the road.

Research has improved the outlook for T1DM over the last decade. Doctors are investigating, for example, how to save insulin-producing cells and extend the honeymoon period as long as possible.

Despite progress towards understanding the science behind T1DM, there remains a significant need to investigate alternative approaches to this disease in order to bring about long-term remission. For this reason, scientists are working hard to develop new treatments that can be given soon after diagnosis to preserve the remaining beta cells.

Currently there is no cure for T1DM; however, with new investigational medications and innovative clinical research studies, such as T1DAL, a new approach towards managing T1DM may be on the horizon.

Enrollees will receive weekly intramuscular injections of alefacept or placebo for two 12 week periods, with a 12-week pause between treatment intervals. This schedule or drug dosing may be altered due to the needs of the subject or at the discretion of the physician investigator.

ELIGIBILITY:
Inclusion Criteria:

* Recent diagnosis (within 100 days of enrollment) of T1DM
* Positive for at least one diabetes autoantibody (Glutamate decarboxylase [GAD-65GAD65], IA2, ZnT8, ICA and Insulin, if obtained within 10 days of the onset of exogenous insulin therapy)
* Peak stimulated C-peptide level > 0.2 pmol/mL following a mixed-meal tolerance test (MMTT)
* Willingness to provide written informed consent (either the subject or the subject's legally authorized representative).

Exclusion Criteria:

* Severe reaction or anaphylaxis to human monoclonal antibodies
* History of malignancy or significant cardiovascular disease (including history of myocardial infarction, angina, use of anti-anginal medicines (e.g., nitroglycerin), or abnormal stress test)
* History of recent or ongoing uncontrolled bacterial, viral, fungal, or other opportunistic infections
* Evidence of infection with hepatitis B virus (HBV) as defined by hepatitis B surface antigen, HBsAg; hepatitis C virus (HCV) defined by anti-HCV antibodies; human immunodeficiency virus (HIV); or toxoplasmosis
* Positive tuberculin skin test (PPD)
* Clinically active infection with Epstein-Barr virus (EBV)-EBV viral load ≥ 10,000 copies per 10^6 PBMCs; cytomegalovirus (CMV) -CMV viral load ≥10,000 copies per mL whole blood; or tuberculosis (TB)
* Diagnosis of liver disease or hepatic enzymes, as defined by ALT and/or AST ≥ 2 times the upper limit of normal
* Prior or current treatment that is known to cause a significant, ongoing change in the course of T1DM or immunologic status, including high-dose inhaled, extensive topical or systemic glucocorticoids
* Current or prior (within the last 30 days) use of metformin, sulfonylureas, glinides, thiazolidinediones, exenatide, liraglutide, DPP-IV inhibitors or amylin
* Current use of any medication known to influence glucose tolerance (e.g., atypical antipsychotics, diphenylhydantoin, thiazide, or other potassium-depleting diuretics, β-adrenergic blockers, niacin)
* Any of the following hematologic abnormalities, confirmed by repeat tests at least 1 week apart:

  1. White blood count <4000/μL or >14,000/μL;
  2. CD4+ count below the lower limit of normal;
  3. Platelet count <150,000 /μL; or
  4. Hemoglobin <10 g/dL.
* Females who are pregnant, lactating, or planning on pregnancy during the 2-year study period
* History of bone marrow transplantation, or autoimmune disease associated with lymphopenia
* Any medical condition that in the opinion of the principal investigator would interfere with safe completion of the trial
* Prior participation in a clinical trial that could potentially affect T1DM or immunologic status
* Receipt of a live vaccine (e.g., varicella, measles, mumps, rubella, cold-attenuated intranasal influenza vaccine, bacillus Calmette-Guérin, and smallpox) in the 6 weeks before enrollment
* Participation in an investigational clinical trial within the last six weeks.

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2011-03; Primary Completion 2013-03 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Rigby, MD, PhD, Principal Investigator — Indiana University
Locations (15):
- United States (15):
  - University of Arizona, Tucson, Arizona
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California - San Francisco, San Francisco, California
  - Barbara Davis Center for Childhood Diabetes - University of Colorado, Aurora, Colorado
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Iowa Hospital & Clinics, Iowa City, Iowa
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Creighton University, Omaha, Nebraska
  - University of North Carolina, Durham, North Carolina
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Participant level data access and additional relevant materials are available to the public in: 1.) the Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts that also provides data analysis tools available to researchers; and 2.) TrialShare, the Immune Tolerance Network (ITN) Clinical Trials Research Portal that makes data from the consortium's clinical trials publicly available.

REFERENCES:
- [Background] Herold KC. Restoring immune balance in type 1 diabetes. Lancet Diabetes Endocrinol. 2013 Dec;1(4):261-3. doi: 10.1016/S2213-8587(13)70123-2. Epub 2013 Sep 23. No abstract available. PMID 24622404
- [Result] Rigby MR, DiMeglio LA, Rendell MS, Felner EI, Dostou JM, Gitelman SE, Patel CM, Griffin KJ, Tsalikian E, Gottlieb PA, Greenbaum CJ, Sherry NA, Moore WV, Monzavi R, Willi SM, Raskin P, Moran A, Russell WE, Pinckney A, Keyes-Elstein L, Howell M, Aggarwal S, Lim N, Phippard D, Nepom GT, McNamara J, Ehlers MR; T1DAL Study Team. Targeting of memory T cells with alefacept in new-onset type 1 diabetes (T1DAL study): 12 month results of a randomised, double-blind, placebo-controlled phase 2 trial. Lancet Diabetes Endocrinol. 2013 Dec;1(4):284-94. doi: 10.1016/S2213-8587(13)70111-6. Epub 2013 Sep 23. PMID 24622414
- [Result] Rigby MR, Harris KM, Pinckney A, DiMeglio LA, Rendell MS, Felner EI, Dostou JM, Gitelman SE, Griffin KJ, Tsalikian E, Gottlieb PA, Greenbaum CJ, Sherry NA, Moore WV, Monzavi R, Willi SM, Raskin P, Keyes-Elstein L, Long SA, Kanaparthi S, Lim N, Phippard D, Soppe CL, Fitzgibbon ML, McNamara J, Nepom GT, Ehlers MR. Alefacept provides sustained clinical and immunological effects in new-onset type 1 diabetes patients. J Clin Invest. 2015 Aug 3;125(8):3285-96. doi: 10.1172/JCI81722. Epub 2015 Jul 20. PMID 26193635
- [Derived] Boyle KD, Keyes-Elstein L, Ehlers MR, McNamara J, Rigby MR, Gitelman SE, Weiner LJ, Much KL, Herold KC. Two- and Four-Hour Tests Differ in Capture of C-Peptide Responses to a Mixed Meal in Type 1 Diabetes. Diabetes Care. 2016 Jun;39(6):e76-8. doi: 10.2337/dc15-2077. Epub 2016 Apr 13. No abstract available. PMID 27208317
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) website — https://www.niddk.nih.gov/
- See also: Immune Tolerance Network (ITN) website — http://www.immunetolerance.org
- See also: Juvenile Diabetes Research Foundation (JDRF) website — http://jdrf.org/about-jdrf/
- Available data/document: Individual Participant Data Set: SDY797 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY797 — ImmPort study identifier is SDY797.
- Available data/document: Study Protocol: SDY797 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY797 — ImmPort study identifier is SDY797. The study protocol is located under the design tab.
- Available data/document: Study summary, -design, -adverse event(s), -demographics, -study files: SDY797 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY797 — ImmPort study identifier is SDY797.ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts. This archive is in support of the NIH mission to share data with the public. Data shared through ImmPort has been provided by NIH-funded programs, other research organizations and individual scientists ensuring these discoveries will be the foundation of future research.
- Available data/document: Individual Participant Data Set: T1DAL ITN045AI — https://www.itntrialshare.org/project/Studies/ITN045AIJCI/Study%20Data/begin.view? — TrialShare study ID is T1DAL ITN045AI.
- Available data/document: Study Protocol: T1DAL ITN045AI — https://www.itntrialshare.org/project/Studies/ITN045AIJCI/Study%20Data/begin.view? — TrialShare study ID is T1DAL ITN045AI.
- Available data/document: Study overview, -data and reports, -schedule of assessments, -study design, -original article & abstracts et al.: T1DAL ITN045AI — https://www.itntrialshare.org/project/Studies/ITN045AIJCI/Study%20Data/begin.view? — TrialShare is a clinical trials research portal developed by the Immune Tolerance Network (ITN) that makes data from the consortium's clinical trials publicly available without charge.Creating an account for ITN TrialShare is free and allows for searching studies of interest.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited during an approximate 84-week accrual period. Initially 66 subjects were planned; however, enrollment ended with 49 subjects as a result of the decision, unrelated to safety reasons, made by Astellas Pharma US, Inc. to discontinue manufacturing Amevive® (alefacept).
Pre-assignment Details: Subjects ages 12 to 35 years who were first diagnosed with type 1 diabetes mellitus (T1DM) within 100 days of enrollment. Subjects were randomly assigned in a 2 to 1 (2:1) ratio to either the alefacept or placebo group.
Groups:
- Alefacept: Subjects in this group received weekly intramuscular injections of alefacept (15 mg) for 2 cycles of 12 weeks each, separated by a 12 week pause in treatment.
Period: Overall Study
Arm/Group | Alefacept | Placebo
Started | 33 | 16
Completed | 31 | 12
Not Completed | 2 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alefacept | Placebo | Total
Number analyzed (Participants) | 33 | 16 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 8 | 25
  Between 18 and 65 years | 16 | 8 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.3 (6.4) | 19.5 (6.2) | 20.0 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 4 | 20
  Male | 17 | 12 | 29
Region of Enrollment [Number; unit: participants]
  United States | 33 | 16 | 49
2-Hour C-peptide Area Under the Curve Result in Response to Standardized Mixed Meal Tolerance Test [Mean (Standard Deviation); unit: pmol/mL] — C-peptide is a substance released by the pancreas into the bloodstream in equal amounts to insulin and reflects how much insulin pancreatic beta cells are making. The MMTT evaluates whether beta cells are producing endogenous insulin. The MMTT was performed in the morning and blood samples for C-peptide collected at baseline (pre-meal) and 15, 30, 60, 90, 120, 150, 180, 210,and 240 minutes post-meal. Results of the stimulated 2-hour post-meal C-peptide AUC are provided. Larger numbers are preferable (better) in these AUC results: more insulin being produced reflects less severe disease.
  pmol/mL | 0.85 (0.42) | 0.64 (0.22) | 0.78 (0.38)

OUTCOME MEASURES:

1. Primary Outcome: 2-Hour C-peptide Area Under the Curve (AUC) Result in Response to Standardized Mixed Meal Tolerance Test (MMTT)
Description: C-peptide is a substance released by the pancreas into the bloodstream in equal amounts to insulin and reflects how much insulin pancreatic beta cells are making. The standardized MMTT evaluates whether beta cells are producing endogenous insulin. The MMTT was performed in the morning and blood samples for C-peptide collected at baseline (pre-meal) and 15, 30, 60, 90, 120, 150, 180, 210,and 240 minutes post-meal. Results of the stimulated 2-hour (e.g., 120 minutes) post-meal C-peptide AUC are provided. Larger numbers are preferable (better) in these AUC results: more insulin being produced reflects less severe disease. C-peptide levels in the serum (e.g., AUC following a standardized MMTT) compared to control group at 1 year post treatment initiation for the evaluation of investigational products intended to preserve endogenous beta-cell function in T1DM trials is recognized by the Center for Drug Evaluation and Research (CDER) at the FDA as a valid efficacy primary endpoint.
Time Frame: Baseline (pre-treatment initiation), Week 52
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: pmol/mL
Arm/Group | Alefacept | Placebo
Number analyzed (Participants) | 33 | 16
pmol/mL
  Baseline (Pre-treatment initiation) | 0.85 (0.42) | 0.64 (0.22)
  Week 52 | 0.86 (0.49) | 0.53 (0.38)
  Change from Baseline(Pre-treatment initiation) | 0.02 (0.27) | -0.12 (0.30)
Statistical Analysis 1: Comparison: Alefacept vs Placebo; Primary imputation method used for missing Month 12 AUC. Measuring range for C-peptide is 0.05-30 ng/mL; Test type: Superiority or Other; p = 0.065, ANCOVA — P-value is for testing treatment effect using an analysis of covariance with baseline ln(AUC+1) as a covariate and change in ln(AUC+1) from baseline as the outcome variable

2. Secondary Outcome: 4-Hour C-peptide Area Under the Curve (AUC) Result in Response to Standardized Mixed Meal Tolerance Test (MMTT)
Description: as for outcome 1
Time Frame: Baseline (Pre-treatment initiation), Week 52, and Week 104
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: pmol/mL
Arm/Group | Alefacept | Placebo
Number analyzed (Participants) | 33 | 16
pmol/mL
  Baseline (Pre-treatment initiation) | 0.84 (0.36) | 0.68 (0.23)
  Week 52 | 0.86 (0.42) | 0.52 (0.35)
  Change from Baseline(Pre-treatment initiation) | 0.02 (0.26) | -0.16 (0.28)
  Week 104 | 0.71 (0.50) | 0.31 (0.30)
  Change from Baseline (Pre-treatment initiation) | -0.13 (0.37) | -0.37 (0.20)
Statistical Analysis 1: Comparison: Alefacept vs Placebo; Primary imputation method used for missing Week 52 AUC. Measuring range for C-peptide is 0.05-30 ng/mL; Test type: Superiority or Other; p = 0.019, ANCOVA — P-value is for testing treatment effect using an analysis of covariance with baseline In(AUC+1) as a covariate and change in In(AUC+1) from baseline as the outcome
Statistical Analysis 2: Comparison: Alefacept vs Placebo; Primary imputation method used for missing Week 104 AUC. Measuring range for C-peptide is 0.05-30 ng/mL; Test type: Superiority or Other; p = 0.002, ANCOVA — [p-value comment as in outcome 2, analysis 1]

3. Secondary Outcome: 2-Hour C-peptide Area Under the Curve (AUC) Result in Response to Standardized Mixed Meal Tolerance Test (MMTT)
Description: as for outcome 1
Time Frame: Baseline (Pre-treatment initiation), Week 52, and Week 104
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: pmol/mL
Arm/Group | Alefacept | Placebo
Number analyzed (Participants) | 33 | 16
pmol/mL
  Baseline (Pre-treatment initiation) | 0.85 (0.42) | 0.64 (0.22)
  Week 52 | 0.86 (0.49) | 0.53 (0.38)
  Change from Baseline(Pre-treatment initiation) | 0.02 (0.27) | -0.12 (0.30)
  Week 104 | 0.66 (0.50) | 0.31 (0.29)
  Change from Baseline (Pre-treatment initiation) | -0.19 (0.34) | -0.33 (0.22)
Statistical Analysis 1: Comparison: Alefacept vs Placebo; Primary imputation method used for missing Week 52 AUC. Measuring range for C-peptide is 0.05-30 ng/mL; Test type: Superiority or Other; p = 0.065, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Alefacept vs Placebo; Primary imputation method used for missing Week 104 AUC. Measuring range for C-peptide is 0.05-30 ng/mL; Test type: Superiority or Other; p = 0.015, ANCOVA — [p-value comment as in outcome 2, analysis 1]

4. Secondary Outcome: Insulin Use in Units Per Kilogram Body Weight Per Day
Description: The need to use insulin is an indication that the body is not producing enough endogenous insulin. Higher amounts of insulin use indicate higher disease activity.
Time Frame: Baseline (Pre-treatment initiation), Week 52, and Week 104
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: Units per day divided by weight in kg
Arm/Group | Alefacept | Placebo
Number analyzed (Participants) | 33 | 16
Units per day divided by weight in kg
  Baseline (Pre-treatment initiation) | 0.33 (0.20) | 0.29 (0.17)
  Week 52 | 0.36 (0.22) | 0.48 (0.27)
  Change from Baseline(Pre-treatment initiation) | 0.02 (0.15) | 0.17 (0.22)
  Week 104 | 0.43 (0.19) | 0.60 (0.24)
  Change from Baseline (Pre-treatment initiation) | 0.10 (0.16) | 0.28 (0.16)
Statistical Analysis 1: Comparison: Alefacept vs Placebo; Week 52 mean insulin use comparison; Test type: Superiority or Other; p = 0.020, ANCOVA — P-value is for testing treatment effect using an analysis of covariance with baseline level as a covariate and change from baseline as the outcome variable
Statistical Analysis 2: Comparison: Alefacept vs Placebo; Week 104 mean insulin use comparison; Test type: Superiority or Other; p = 0.002, ANCOVA — [p-value comment as in outcome 4, analysis 1]

5. Secondary Outcome: Major Hypoglycemic Events Occurring From Randomization
Description: Major hypoglycemic events are defined as a glucose concentration <55 mg/dL (grades 2-5, NCI-CTCAE version 3.0), or clinically: involving seizure(s) or involving loss of consciousness (coma), or requiring assistance from another individual in order to recover.
Time Frame: Baseline to Week 52 and Week 52 to Week 104
Population: Intent-to-treat
Measure: Number; unit: Major Hypoglycemic Events
Arm/Group | Alefacept | Placebo
Number analyzed (Participants) | 33 | 16
Major Hypoglycemic Events
  Baseline to Week 52 | 357 | 274
  Week 52 to Week 104 | 252 | 251
Statistical Analysis 1: Comparison: Alefacept vs Placebo; Hypoglycemic Events Occurring from Baseline to Week 52; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value is from a poisson regression comparing the person-year adjusted event rates between the two treatment groups
Statistical Analysis 2: Comparison: Alefacept vs Placebo; Hypoglycemic Events Occurring from Week 52 to Week 104; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value is from a poisson regression comparing the person-year adjusted event rates between the two treatment groups

6. Secondary Outcome: Hemoglobin A1c
Description: Glycosylated hemoglobin (HbA1c) is a measure of the average plasma concentration of blood sugar (glucose) over the previous three months and measures the level of optimal management of underlying disease. An HbA1c level of 5.6% or less is considered normal. HbA1c levels of 6.5% or higher is typical for individuals with Type 1 Diabetes Mellitus (T1DM). The closer HbA1c levels are to normal, the better controlled the disease is.
Time Frame: Baseline (Pre-treatment initiation), Week 52, and Week 104
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: HgbA1c percent (%)
Arm/Group | Alefacept | Placebo
Number analyzed (Participants) | 33 | 16
HgbA1c percent (%)
  Baseline (Pre-treatment initiation) | 7.2 (1.5) | 7.1 (1.5)
  Week 52 | 6.9 (1.9) | 7.2 (1.3)
  Change from Baseline(Pre-treatment initiation) | -0.1 (1.4) | 0.0 (1.3)
  Week 104 | 7.4 (1.6) | 7.5 (1.3)
  Change from Baseline (Pre-treatment initiation) | 0.4 (1.5) | 0.3 (1.2)
Statistical Analysis 1: Comparison: Alefacept vs Placebo; Week 52 mean HbA1C comparison; Test type: Superiority or Other; p = 0.746, ANCOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Alefacept vs Placebo; Week 104 mean HbA1C comparison; Test type: Superiority or Other; p = 0.942, ANCOVA — [p-value comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: Enrollment through participant's last visit, up to Week 104
Arm/Group | Alefacept | Placebo
Serious Adverse Events (participants affected / at risk) | 1/33 | 0/16
Other Adverse Events (participants affected / at risk) | 33/33 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alefacept (N=33) | Placebo (N=16)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alefacept (N=33) | Placebo (N=16)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 4 (13) | 2 (8)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 1 (1)
Episcleritis (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (8) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 2 (3)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (8) | 4 (5)
Toothache (Gastrointestinal disorders) | 2 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (6) | 2 (2)
Chills (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 4 (5) | 1 (1)
Influenza like illness (General disorders) | 2 (7) | 2 (3)
Pain (General disorders) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 3 (3) | 2 (3)
Allergy to arthropod bite (Immune system disorders) | 2 (2) | 0 (0)
Seasonal allergy (Immune system disorders) | 4 (4) | 2 (3)
Ear infection (Infections and infestations) | 2 (2) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 4 (4) | 2 (5)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 2 (2)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 9 (16) | 3 (4)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 6 (7) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 1 (2)
Rash pustular (Infections and infestations) | 2 (2) | 0 (0)
Rhinitis (Infections and infestations) | 2 (4) | 0 (0)
Sinusitis (Infections and infestations) | 6 (9) | 3 (9)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 19 (40) | 7 (14)
Viral infection (Infections and infestations) | 3 (4) | 2 (2)
Vulvovaginal candidiasis (Infections and infestations) | 2 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 6 (6) | 4 (5)
Excoriation (Injury, poisoning and procedural complications) | 4 (5) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Nail avulsion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 7 (14) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 6 (8) | 2 (4)
CD4 lymphocytes decreased (Investigations) | 2 (6) | 0 (0)
Cardiac murmur (Investigations) | 3 (3) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Low density lipoprotein increased (Investigations) | 2 (2) | 0 (0)
Neutrophil count abnormal (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 3 (3) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 30 (600) | 15 (516)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (7) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (9)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 14 (32) | 5 (9)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Muscle contractions involuntary (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 1 (2)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 2 (3)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 2 (2)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 4 (6) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (4)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (2)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Enrollment ended early with 49 subjects (instead of the planned 66) as a result of the decision, unrelated to safety reasons, made by Astellas Pharma US, Inc. to discontinue manufacturing Amevive® (alefacept).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No